CLINICAL TRIAL: NCT04453033
Title: Double-blind, Randomized Controlled Trial to Demonstrate Efficacy of Celeste® Specialized Phototherapy in Treating Parkinson's Disease.
Brief Title: DB RCT for Specialized Phototherapy in Parkinson's Disease.
Acronym: LIGHT-PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PhotoPharmics, Inc. (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-2401
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a six-month, randomized, double-blind, controlled, parallel group study with visits at screening, baseline, weeks 13 and 26, and blinded coordinator calls throughout the study for safety and efficacy assessments. This study will use a remote trial design, which will allow participants to be recruited nationally and evaluated centrally using video conferencing. All study participants will have their eligibility assessed and confirmed by a study coordinator and a PD specialist (primary investigator). Participants will complete the secondary outcome measures, which are Patient Response Outcomes (PRO's), and will be assisted by a blinded coordinator to ensure completeness of answers. A blinded rater will conduct the Primary Outcome Measure as well as the MDS-UPDRS. All assessments will be conducted by video at Baseline, Week 13, and Week 26 visits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research suggests that certain wavelengths of light are more effective in treating Parkinson's, which means this therapeutic light device does not need to be nearly as bright as traditional light therapy. This study will test a light therapy device (Celeste® specialized light therapy device). We are testing two devices in this study: an active device which has these special wavelengths, and a control device which does not have the special wavelengths. Both lights look the same, and it is not possible to tell which light has the effective wavelength by looking at it. No one involved in the study (patients, families, doctors, investigative staff) knows which type of light therapy each person receives. A Device Technician, separate from the trial, will assist the participants in the device setup. Participants will be instructed not to disclose any aspects of their device. All study staff will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Investigational Device (Active Comparator): The Celeste device resembles a large tablet. It has a protective cover that folds into a stand and is magnetically attached to the back of the device. It produces a low intensity of specific bandwidths of light believed to be responsible for circadian and alerting responses in humans. The overall emission produces a pleasing soft glow of light.
  Interventions: Device: Celeste Specialized Phototherapy Device
- Control Device (Sham Comparator): The Control device is identical in appearance to Celeste. When turned on, the device emits a soft diffused light that is indistinguishable in color from the Active Device. However, this device produces a different amount of the specific wavelengths thought to be effective in the Active Device. It is impossible to tell the difference between the sham device and the active device by looking at them.
  Interventions: Device: Celeste Specialized Phototherapy Device

INTERVENTIONS:
Device: Celeste Specialized Phototherapy Device — Ocular phototherapy light panel

SUMMARY:
This is a pivotal study to determine whether light therapy can improve non-motor and motor function in Parkinson's disease, on top of current best medical treatment.

DETAILED DESCRIPTION:
Six month double blind, randomized controlled study with virtual clinic visits at baseline, week 13 and week 26. The Celeste specialized phototherapy device is similar to a tablet with a stand that allows the device to be angled towards the participant's face. The light is to be used each evening in the home for 1 hour, while the participant watches TV, eats dinner, reads, etc. The primary outcome measure is the Parkinson's Disease Questionnaire-39 Summary Index (PDQ-39SI). The PDQ-39 is a patient-reported, quality of life scale. The key secondary endpoint is Parts 1 and 2 of the Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS). The MDS-UPDRS Parts 1 and 2 measure non-motor and motor function in Parkinson's. Participants will be assessed via online videoconferences.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Parkinson's disease as determined by the study PI, in keeping with the UK PD Society Brain Bank Criteria for the Diagnosis of PD

Responsiveness to dopaminergic medication, as judged by the rater, and have been using treatment for at least the past 1 year

Relatively good eyesight as attested to by participants (Corrective lenses of at least 20/60)

Stable levodopa and other anti-PD medications for at least 28 days prior to screening -

Exclusion Criteria:

Diagnosis of an atypical Parkinsonian syndrome

Significant OFF state or bothersome dyskinesias that in the judgment of the rater, would interfere with participation in the study.

An anticipated need for a change in dopamine replacement therapy, concomitant medications, OTC/supplements, or other alternative therapies during the participant's involvement in the investigation

History of previous light therapy use for PD

-

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Questionnaire-39 (PDQ-39) | 26 weeks
  The Parkinson's Disease Questionnaire-39 (PDQ-39) is a patient-reported rating scale for quality of life in Parkinson's disease. Respondents affirm if they have experienced problems due to their disease using a five point scale from never (0 points) to always (4 points, or worse) in doing common activities. The PDQ-39 is comprised of 8 domains: mobility, emotion, activities of daily living, cognition, stigma, social support, communication, bodily discomfort. Total possible range of scores = 0 - 156, with higher scores representing worse severity.

SECONDARY OUTCOMES:
Movement Disorders Society-Unified Parkinson's Disease Rating Scale, Sum or Parts 1+2 | 26 weeks
  MDS-UPDRS Part 1: Non-motor impact of experiences of daily living. Part I has 13 questions, the first 6 are assessed by the examiner, and the remaining 7 are usually self assessed, but may include the patient's caregiver. Each question = 0-4, range= 0 - 65, with higher scores representing worse severity.
  MDS-UPDRS Part II: Motor Aspects of Experiences of Daily Living: This portion of the scale assesses the motor impact of PD on patients' experiences of daily living. There are 13 questions which are a component of the self-administered Patient Questionnaire. Each question = 0-4, range = 0-65. with higher scores representing worse severity.

OTHER OUTCOMES:
Parkinson's Disease Health Index (PD-HI) | 26 weeks
  The Parkinson's Disease Health Index (PD-HI) is a highly sensitive disease specific patient response outcome measure, designed to measure the longitudinal progression of Parkinson's disease and treatment effectiveness. The PD-HI combines 13 sub-domains according to the prevalence and impact of Parkinson's symptoms on patients. Each domain is ranked by the individual on a Likert scale of 0-100, according to how the domain is currently affecting them. A higher score reflects a more severe condition. An algorithm is used to compute the total score, with 100 being the highest score possible. The PD-HI will be used at Baseline, at Week 13, and at Week 26.
Epworth Sleepiness Scale (ESS) | 26 weeks
  The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness to help in diagnosing sleep disorders. The ESS questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 (none) to 3 (worse) for eight different everyday situations. The total range is 0 - 24, with higher scores representing worse severity.
Scales for Outcomes in Parkinson's Disease - Sleep (SCOPA-Sleep) | 26 weeks
  The SCOPA-SLEEP is a frequency measure scale to assess the character and quantify the various aspects of sleep problems in Parkinson's disease. The SCOPA-Sleep consists of 13 items, including information about the use of sleeping tablets. Questions range from 0 to 4 in severity, (Question 7, Quality of Sleep, ranges from 0-7). A higher total score indicates more severe sleep problems.
Beck Depression Inventory -II (BDI-II) | 26 weeks
  The Beck Depression Inventory (BDI) is a 21-question multiple choice inventory to measure the severity of depression. Each question is scored on a scale value of 0 to 3. The cutoffs used are: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; and 29-63: severe depression. Higher total scores indicate more severe depressive symptoms.
Beck Anxiety Scale (BAI) | 26 weeks
  The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63). Input from a caregiver to the participant is acceptable.
Montreal Cognitive Assessment (MoCA) | 26 weeks
  The Montreal Cognitive Assessment (MoCA) is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The MoCA will be used at screening, mainly for characterization purposes and to assist the site investigators in their decisions to include participants in the trial. Higher scores indicate better cognitive function, while a score below 26 may indicate mild cognitive impairment. The MoCA will be assessed at baseline, Week 13, and Week 26.
Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part 3 (Modified) | 26 weeks
  The MDS-UPDRS Part 3 is the motor examination section of the MDS-UPDRS. It is completed by the Evaluator. Part 3 evaluates speech, tremor, bradykinesia, rigidity, spontaneity of movement, gait, and balance. Because rigidity (3.3) and postural stability (3.12) cannot be measured remotely, a modified version, which omits these questions will be used. The same rater will evaluate the same participants whenever possible, and at the same time of day. Raters must be certified in the use of the MDS-UPDRS.
EuroQol-5 Dimensions (EQ-5D-5L) | 26 weeks
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D is a standardized measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. The instrument comprises a short descriptive system questionnaire covering five areas which assess quality of life issues, and a visual analogue scale (EQ VAS) that provides a simple descriptive profile of a respondent's health state. The 5L refers to five levels (0-4) of increasing severity for each question.
Parkinson's Disease Patient Report of Problems (PD PROP) | 26 Weeks
  The Parkinson's Disease Patient Report of Problems is an online assessment tool that allows patients to describe their most bothersome problems and how these problems affect their daily functioning in their own terms. The tool then uses algorithms and machine learning to quantify those problems and their progression with greater sensitivity and detail that is unavailable from other assessments. The PD-PROP classifies these answers into a total of 56 clinically meaningful symptoms, representing four motor and six non-motor domains. The PD PROP will be assessed at baseline, Week 13, and Week 26.

CONTACTS AND LOCATIONS:
Overall Officials: Ray Dorsey, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
In addition to submitting the study design and results to www.clinicaltrials.gov, the final results of the study will be published in a peer-reviewed journal after the generation of the clinical study report. Subsequent to publication and FDA submission, PhotoPharmics intends to make the data available to qualified researchers for collaboration. The general results of the trial may also be made available to study participants during a webinar.